CLINICAL TRIAL: NCT05246865
Title: The Role of 11-oxygenated Androgens in Androgen Excess and Metabolic Dysfunction of Women With Polycystic Ovary Syndrome
Brief Title: Impact of 11-oxygenated Androgens on Metabolic Dysfunction of Women With Polycystic Ovary Syndrome
Acronym: 11OXO-PCOS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: RG_19-038
Record Dates: First submitted 2019-07-26; First posted 2022-02-18 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-11

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Dehydroepiandrosterone; adrenosterone

STUDY DESIGN:
Intervention Model Description: A prospective human in-vivo physiology study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Women with PCOS (Experimental): Women with polycystic ovary syndrome
  Interventions: Drug: oral androgen challenge with dehydroepiandrosterone (DHEA)
- Age and BMI-matched healthy volunteers (Experimental): Otherwise healthy women without PCOS but matching in age and body mass index to the above group
  Interventions: Drug: oral androgen challenge with dehydroepiandrosterone (DHEA)

INTERVENTIONS:
Drug: oral androgen challenge with dehydroepiandrosterone (DHEA) — The oral androgen challenge is a safe and well-validated means of studying the androgen generation profiles of different study groups.
  Other Names: oral androgen challenge with 11-ketoandrostenedione

SUMMARY:
Polycystic ovary syndrome (PCOS) affects 10% of all women and usually presents with irregular menstrual periods and difficulties conceiving. It is also a lifelong metabolic disorder and affected women have an increased risk of type 2 diabetes, high blood pressure, and heart disease. Increased blood levels of male hormones, also termed androgens, are found in most PCOS patients. Androgen excess appears to impair the ability of the body to respond to the sugar-regulating hormone insulin (also termed 'insulin resistance'). Androgens circulating in the blood in women with PCOS are comprised of classic androgens (for example testosterone), and the less-characterised 11-oxygenated androgen subclass that arises from the adrenal glands. The investigators have recently demonstrated that 11-oxygenated androgens make up the majority of circulating androgens in women with PCOS.

In preliminary studies using minimally invasive adipose tissue sampling, the investigators have found that the fat tissue of women with PCOS overproduces classic androgens. This can lead directly to disturbances in the ability of fat cells to store fat effectively (lipotoxicity), resulting in insulin resistance and the consequent risk of liver damage. However, there are no published studies on in vivo androgen concentrations in the adipose tissue of women with PCOS. Furthermore, the scientific community do not have any information on whether adipose concentrations of 11-oxygenated androgens are also increased in women with PCOS.

Research Questions The investigators aim to examine the metabolism of classic and 11-oxygenated androgens in detail in both circulations and in the adipose tissue of women with PCOS. The investigators will examine how precursor variants of both 11-oxygenated and classic androgens, which are converted by the body into active hormones, are broken down (metabolised) within the adipose tissue of women with PCOS. The investigators will also investigate if the 11-oxygenated androgens have a differential impact on metabolic function as compared to classic androgens. This will give important insights into the adipose tissue metabolome in women with PCOS, and how locally generated androgens impact on adipose tissue function and metabolic risk.

DETAILED DESCRIPTION:
In part A of the study, women with PCOS and obesity, identified from the previously established DAISy-PCOS cohort, and age- and BMI-matched healthy volunteers identified by advertisements, will be invited for a screening visit (Visit 1) at the National Institute of Health Research-Wellcome Trust Clinical Research Facility at the Queen Elizabeth Hospital Birmingham. Once eligibility (described in detail in Section 7.1) has been confirmed, a written informed consent will be obtained, and the volunteers will be invited to three further metabolic assessment visits after an overnight fast.

While Visits 2 and 3 (Study days 1 and 2, respectively) will be for the assessment of responses to an androgen-precursor challenge, Visit 4 (Study day 3) will run in the same format as the previous two Study days except no androgen will be administered. During each visit, study participants will undergo abdominal adipose tissue vein cannulation, whereby a catheter will be inserted (under ultrasound guidance and with local anaesthetic) into one of the veins of the abdominal fat tissue. Ultrasound Doppler and ethanol dilution by microdialysis will be employed to assess adipose tissue blood flow. A further catheter will be inserted into a vein on the back of the hand which will be placed a hot air box in order to obtain arterialised blood. Finally, a catheter will be inserted into an antecubital vein for the purposes of stable isotope infusion. Blood samples from the hand vein and from the abdominal adipose tissue vein will be taken in tandem every 30 minutes for measurement of various metabolites, androgens, and non-targeted metabolome studies. Salivary samples will be collected every 30 minutes in the first hour and hourly thereafter until the end of the study. Urine will be collected throughout the Study Visit. At time point 240 min, a standardised high-fat meal containing palmitate labelled with a stable isotope will be given to the participant, and measurements will continue, to assess how their metabolism responds to the meal. Furthermore, fat tissue biopsies will be taken from the subcutaneous abdominal adipose tissue at the end of each study day. These fat biopsies will undergo RNA extraction for transcriptional profiling by RNA-sequencing and will be used for tissue incubation to determine their androgen-generating and metabolic capacity.

On Visits 2 and 3, participants will be administered either the classic androgen pathway precursor dehydroepiandrosterone or the 11-oxygenated androgen pathway precursor 11-ketoandrostenedione at time point 0 min. No androgen precursors will be administered during Visit 4. Otherwise, Visits 2-4 will be identical in their flow.

In part B of the study, paired subcutaneous and omental adipose tissue samples (up to 5 g), as well as a blood sample, are collected from female volunteers undergoing elective abdominal surgery. These tissue samples alongside the subcutaneous tissue obtained from the in vivo study (part A) will be used for ex vivo incubations with androgen precursors to study androgen activation and its metabolic impact. Additionally, the effect of Aldo-Keto Reductase Family 1 Member C3 inhibition on androgen activation will be assessed in ex vivo incubations. After the incubation, the culture medium and/or the tissue will be used for metabolome analysis (non-targeted global metabolome and steroid metabolome profiling) and transcriptome analysis. The blood sample will be used for serum multi-steroid profiling.

ELIGIBILITY:
Part A

Inclusion Criteria:

* BMI between 30-40 kg/m2
* Age range 18-40 years
* Ability to provide informed consent

For women participating in the PCOS group, the diagnosis of PCOS will be established during their recruitment to DAISy-PCOS study on the basis of the Rotterdam Consensus Criteria for the Diagnosis of PCOS, as recommended by the current international PCOS guidelines (at least 2 out of 3 criteria):

* Androgen excess (clinical and/or biochemical evidence)
* Chronic oligo-/anovulation (clinical and/or biochemical evidence)
* Polycystic appearance of the ovaries on ultrasound (according to the most recent guidelines (10), taking into account the higher resolution capacity of modern ultrasound, the presence of ovarian PCOS morphology is defined as follows: 20 or more follicles of 2-9mm in diameter and/or an increased ovarian volume >10 millilitre [without a cyst or dominant follicle] in either ovary) In addition, we will perform clinical and/or biochemical exclusion, as appropriate, of other conditions that could explain the above manifestation (e.g. congenital adrenal hyperplasia, Cushing's syndrome, Prolactinoma, adrenal and gonadal tumours)

Exclusion Criteria:

* Pregnancy or breastfeeding at the time of planned recruitment
* History of significant renal (eGFR<30) or hepatic impairment (aspartate aminotransferase or alanine transaminase >two-fold above ULN; pre-existing bilirubinaemia >1.2 ULN)
* Any other significant disease or disorder that, in the opinion of the Investigator, may either put the participant at risk because of participation in the study, or may influence the result of the study, or the participant's ability to participate in the study.
* Participants who have participated in another research study involving an investigational medicinal product in the 12 weeks preceding the planned recruitment
* Glucocorticoid use via any route within the last six months
* Current intake of drugs known to impact upon steroid synthesis or metabolism or on metabolic function or intake of such drugs during the six months preceding the planned recruitment
* Use of oral or transdermal hormonal contraception in the three months preceding the planned recruitment
* Use of contraceptive implants in the twelve months preceding the planned recruitment
* Allergy or intolerance to any of the ingredients in the high fat meal, or any of the ingredients in the dehydroepiandrosterone and 11-ketoandrostenedione preparations.
* Diabetes or impaired glucose metabolism

Part B Inclusion criteria

* Women undergoing elective, abdominal, non-cancer surgery
* Age range 18-70 years
* Ability to provide informed consent

Exclusion criteria

* Pregnancy or breastfeeding at the time of planned recruitment
* Glucocorticoid use via any route within the last six months
* Current intake of drugs known to impact upon steroid synthesis or metabolism or on metabolic function or intake of such drugs during the six months preceding the planned recruitment
* Type 1 diabetes
* Medical treatment of type 2 diabetes

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-10-10 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2025-05-30 (Estimated)

PRIMARY OUTCOMES:
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline height | 3 years
  During Visit 1, the research team will measure height in centimetres
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline weight | 3 years
  During Visit 1, the research team will measure weight in kilogram
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline body mass index (BMI) | 3 years
  During Visit 1, weight and height will be combined to report BMI in kg/m^2
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline waist circumference | 3 years
  During Visit 1, the research team will measure Waist circumference to nearest centimetre
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline blood pressure | 3 years
  During Visit 1, the research team will measure both systolic and diastolic Blood pressure in mmHg after 10 minutes in sitting position
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline urea & electrolytes | 3 years
  During Visit 1, the research team will collect blood to measure urea & electrolytes in mmol/L
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline liver function test | 3 years
  During Visit 1, the research team will collect blood to measure liver function tests in mmol/L
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline haemoglobin | 3 years
  During Visit 1, the research team will collect blood to measure haemoglobin in grams per litre
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline white cell and platelet count | 3 years
  During Visit 1, the research team will collect blood to measure White cell and platelets in number of cells per ml
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline lipid profile | 3 years
  During Visit 1, the research team will collect blood to measure lipid profile in mmol/L
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline glucose | 3 years
  During Visit 1, the research team will collect blood to measure glucose in mmol/L
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline glycated haemoglobin | 3 years
  During Visit 1, the research team will collect blood to measure glycated haemoglobin (HbA1c) in mmol/mol
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline thyroid function test | 3 years
  During Visit 1, the research team will collect blood to measure thyroid function test in mIU/L
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline Dehydroepiandrosterone (DHEAS) | 3 years
  During Visit 1, the research team will collect blood to measure DHEAS in µmol/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline androstenedione | 3 years
  During Visit 1, the research team will collect blood to measure androstenedione in µmol/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline testosterone | 3 years
  During Visit 1, the research team will collect blood to measure testosterone in nmol/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline sex hormone binding globulin | 3 years
  During Visit 1, the research team will collect blood to measure sex hormone binding globulin in nmol/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline 17-hydroxyprogesterone | 3 years
  During Visit 1, the research team will collect blood to measure 17-hydroxyprogesterone in nmol/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline prolactin | 3 years
  During Visit 1, the research team will collect blood to measure prolactin in mIU/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline Follicle-stimulating hormone | 3 years
  During Visit 1, the research team will collect blood to measure Follicle-stimulating hormone in IU/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline luteinizing hormone | 3 years
  During Visit 1, the research team will collect blood to measure luteinizing hormone in IU/L
overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline oestradiol | 3 years
  During Visit 1, the research team will collect approx 20 ml of blood to measure oestradiol in pmol/L.
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-understanding steroidal activity in peripheral blood mononuclear cells. | 3 years
  During Visit 1, the research team will collect approx 63 ml of blood to extract peripheral blood mononuclear cells for further experiments to measure the impact of classic and 11-oxygenated androgen precursors on downstream steroid profile
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism- to study the changes in steroid levels over time in arterialized hand vein | 3 years
  Visit 2 to 4, the research team will collect blood samples (1-2ml each time) from arterialized hand vein to study the changes in steroid levels from -90 to 480 min at 30 min intervals
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism- to study the changes in steroid levels over time in abdominal vein | 3 years
  Visit 2 to 4, the research team will collect blood samples (1-2ml each time) from abdominal vein to study the changes in steroid levels from -90 to 480 min at 30 min intervals
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism to study the changes in salivary steroid levels over time | 3 years
  Visit 2 to 4, the research team will collect salivary samples (1-2ml each time) to study the changes in steroid levels at 0, 30, and 60 minutes and hourly thereafter until the end of Study Visits.
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-to study the changes in urinary steroid levels over time | 3 years
  Visit 2 to 4, the research team will collect urine from time point 0 to 480 minutes to study the changes in steroid levels
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism-establishing baseline hormone levels for part B of the study | 3 years
  for Part B of the study, a blood sample (approx 7 ml) is collected from female volunteers undergoing elective abdominal surgery to establish baseline hormonal levels
The impact of classic and 11-oxygenated androgen precursors on systemic circulation of overall steroid profile and its impact on lipid and glucose metabolism- to study the downstream conversion of steroid precursor in omental and subcutaneous fat | 3 years
  for Part B of the study, paired subcutaneous and omental adipose tissue samples (up to 5 g) are collected from female volunteers undergoing elective abdominal surgery.
  * the concentration of classic and 11-oxygenated androgen metabolites (androstenedione, testosterone, dihydrotestosterone, 11-ketoandrostenedione, 11-hydroxyandrostenedione, 11-ketotestosterone, 11-hydroxytestosterone) will be measured in the culture medium by liquid chromatography tandem mass spectrometery in nmol/L.
  * the relative abundance of all detectable metabolites will be determined by untargeted metabolomics using liquid chromatography tandem mass spectrometery.
  * the tissue will be used for gene expression analysis: Quantitative PCR will be used to determination of the relative abundance of specific mRNA transcripts. RNAseq will be used to quantify the abundace of all mRNA transcripts of the transciptome.

CONTACTS AND LOCATIONS:
Overall Officials: Wiebke Arlt, Dsc, Principal Investigator — Director, Institute of Metabolism and Systems Research (IMSR)
Locations (1):
- Institute of Metabolism and Systems Research, Birmingham, West Midlands, United Kingdom